CLINICAL TRIAL: NCT03135769
Title: A Phase II Trial of Avelumab in Chemo-resistant Gestational Trophoblastic Neoplasias (GTN)
Brief Title: Avelumab in Chemo-resistant Gestational Trophoblastic Neoplasias
Acronym: TROPHIMMUN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL16_0123
Record Dates: First submitted 2017-04-06; First posted 2017-05-01 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Gestational Trophoblastic Neoplasias (GTN)
Keywords: avelumab; PDL1; Gestational Trophoblastic Neoplasias; GTN; Hydatiform mole; hCG

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Avelumab (Experimental): Avelumab administration at 10 mg/kg every 14 days during 6 months maximum
  Interventions: Drug: Avelumab administration at 10mg/kg

INTERVENTIONS:
Drug: Avelumab administration at 10mg/kg — Avelumab administration at 10 mg/kg as a 1 hour IV infusion once every 14 days during 6 months (maximum).

SUMMARY:
Gestational trophoblastic neoplasias (GTN) are characterized by the persistence of elevated hCG titers after complete uterine evacuation of a partial hydatidiform mole (PHM) or a complete hydatidiform mole. GTN patients are commonly treated with single agent treatment (methotrexate or actinomycine-D) or polychemotherapy (first line treatment EMA-CO) according to the predicted risk of resistance to single agent treatment by FIGO score. GTN patients with resistance to these treatments are treated with another single agent drug or polychemotherapy regimens.

Chemotherapy standard regimens are old and toxic for these young lady patients, with potential long term effects detrimental for further maternity and quality of life. There is a need for modern targeted agents with better benefit/toxicity profiles.

There is a strong rational for investigating the anti-PDL1 monoclonal antibody avelumab in chemoresistant GTN patients. Several elements suggest that the normal pregnancy immune tolerance is "hijacked" by GTN cell for proliferating :

* Spontaneous regressions of metastasic GTN are regularly observed, thereby the role of immune system for rejecting GTN cells.
* Strong and constant overexpression of PDL1 and NK cells has been found in all subtypes and settings of GTN tumors from French reference gestational trophoblastic center.
* The case of complete and durable response to pembrolizumab was reported in a patient with multi chemo-resistant GTN.

ELIGIBILITY:
Inclusion criteria for all patients :

* Woman older than 18 years - Patients with Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Patients with adequate bone marrow function :

  * Absolute neutrophil granulocyte count ≥ 1.5 x 10 9 /L
  * Platelet count ≥ 100 x 10 9 /L
  * Haemoglobin ≥ 9.0 g/dL (may have been blood transfused).
* Patients with adequate renal function :

  * Calculated creatinine clearance >= 30 ml/min according to the Cockcroft-Gault formula (or local institutional standard method)
* Patients with adequate hepatic function

  * Serum bilirubin ≤ 1.5 x UNL and AST/ALT ≤ 2.5 X UNL (≤ 5 X UNL for patients with liver metastases)
* Patients must have a life expectancy ≥ 16 weeks
* Confirmation of non-childbearing status for women of childbearing potential. An evolutive pregnancy can be ruled out in the following cases:

  * in case of a previous hysterectomy
  * if serum hCG level ≥ 2 000 IU/L and no intra or extra-uterine gestational sac is detected on pelvic ultrasound
  * if serum hCG level < 2 000 IU/L on a first measurement and serum hCG increases <100% on a second measurement performed 3 days later
* Highly effective contraception if the risk of conception exists. (Note: The effects of the trial drug on the developing human fetus are unknown; thus, women of childbearing potential must agree to use 2 highly effective contraceptions, defined as methods with a failure rate of less than 1 % per year. Highly effective contraception is required at least 28 days prior, throughout and for at least 60 days after avelumab treatment.
* Patients who gave their written informed consent to participate in the study
* Patients affiliated to a social insurance regime
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Cohort A specific inclusion criteria :

- Patients with gestational trophoblastic disease resistant to mono-chemotherapy (methotrexate and/or actinomycine-D

Cohort B specific inclusion criteria :

* Patients with gestational trophoblastic disease resistant to polychemotherapy (such as EMA-CO; EMA-EP; BEP; … regimens) without limitation in the number of previous chemotherapy lines
* Patients with limited risk of fast progression, according to "Centre de reference des maladies trophoblastiques". In the case where a validated therapeutic alternative is available (platinum salt-based chemotherapy in case of resistance to polychemotherapy without platinum salt), the patient must have been informed and the therapeutic alternative will be proposed in priority.

Exclusion Criteria:

* Prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti- CTLA 4 (including ipilimumab, tremelimumab or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways).
* Illness, incompatible with avelumab, such as congestive heart failure; respiratory distress; liver failure; allergy.
* Patients with second primary cancer, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for ≥ 5 years.
* All subjects with brain metastases, except those meeting the following criteria:

  * Brain metastases that have been treated locally and are clinically stable for at least 2 weeks prior to enrollment
  * No on-going neurological symptoms that are related to the brain localization of the disease (sequelae that are a consequence of the treatment of the brain metastases are acceptable)
  * Subjects with brain metastases must be either off steroids except a stable or decreasing dose of <10mg daily prednisone (or equivalent)
* Patients receiving any systemic chemotherapy, radiotherapy (except for palliative reasons), within 2 weeks from the last dose prior to study treatment (or a longer period depending on the defined characteristics of the agents used). The patient can receive a stable dose of bisphosphonates for bone metastases, before and during the study as long as these were started at least 4 weeks prior to treatment with study drug.
* Persistent toxicities (>CTCAE grade 1) with the exception of alopecia and sensory neuropathy ≤ grade 2, caused by previous cancer therapy.
* Treatment with other investigational agents
* Bowel occlusive syndrome, inflammatory bowel disease, immune colitis or other gastro-intestinal disorder that does not allow oral medication such as malabsorption.
* Clinically significant (i.e active) cardiovascular disease : cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication
* Patients with severe acute or chronic medical conditions including immune pneumonitis, inflammatory bowel disease, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
* Known severe hypersensitivity reactions to monoclonal antibodies, any history of anaphylaxis, or uncontrolled asthma (ie, 3 or more features of partially controlled asthma Global Initiative for Asthma 2011).
* Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS) related illness.
* Active infection requiring systemic therapy.
* Positive test for HBV surface antigen and / or confirmatory HCV RNA (if anti-HCV antibody tested positive)
* Administration of a live vaccine within 4 weeks prior the first dose of avelumab.
* Treatment with oral anticoagulant such Coumadin.
* Current or prior use of immunosuppressive medication within 7 days prior to start of study treatment. The following are exceptions to this exclusion criterion:

  * Intranasal, inhaled, topical steroids, or local steroid injections (eg, intra-articular injection);
  * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or equivalent;
  * Steroids as premedication for hypersensitivity reactions (eg, CT scan premedication).
* Active autoimmune disease that might deteriorate when receiving an immunostimulatory agents. Patients with diabetes type I, vitiligo, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible.
* Female patients who are pregnant or lactating, or are of childbearing potential and not practicing a medically acceptable method of birth control
* Resting ECG with QTc > 470msec on 2 or more time points within a 24 hour period or family history of long QT syndrome.
* Prior organ transplantation, including allogeneic stem cell transplantation (excluding autologous bone marrow transplant)
* Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE Grade ≥ 3)
* Patients under guardianship.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2020-12-02 (Actual); Study Completion 2021-03-17 (Actual)

PRIMARY OUTCOMES:
The rate of patients with successful normalization of hCG assays | up to 6 months
  Clinical efficacy of avelumab administration will be evaluated by the rate of patients with successful normalization of hCG assays allowing for treatment discontinuation (hCG normalization). Patients will continue on treatment until the hCG assays, measured weekly, reach the institutional normal threshold and then for 3 additional cycles.

SECONDARY OUTCOMES:
Resistance free survival | up to 6 months
  Number of patients alive free resistance (defined as a rise ≥ 20% rise over between two assays in three consecutive weekly hCG assays or plateau ≤ 10% decrease between two assays in four consecutive weekly hCG)
Progression free survival | up to 6 months
  Number of patients alive progression free survival (defined as a rise ≥ 20% rise over between two assays in three consecutive weekly hCG assays or plateau ≤ 10% decrease between two assays in four consecutive weekly hCG)
Overall survival | up to 6 months
  Number of patients alive 1 months after the end of treatment.
Overall response rate according to RECIST | up to 6 months
  Radiological response to avelumab assessed by the overall response rate according to RECIST version 1.1 criteria and immune-related RECIST criteria assessed by imaging (TAP CT scanner and / or MRI if contraindication) after cycle 4, 8 and 12
NCI CTCAE version 4.0 | up to 7 months
  The safety of avelumab administration will be evaluated throughout the duration of treatment (6 months max) and until the end of patient follow up (1 month after treatment discontinuation) according to NCI CTCAE version 4.0
Kinetics of hCG | up to 7 months
  Modeled hCGres parameter calculated with weekly values of hCG measured during treatment days after start of Avelumab treatment.
PD-L1 expression in tumor samples | up to 7 months
  To predict the efficacy of anti-PD-L1 immunotherapy, we will quantify and characterize the intra and peritumoral immune infiltrate of GTN
Phenotype of the intratumoral immune cell infiltrate | up to 7 months
  Immunohistochemistry with anti PD-L1, anti CD3, anti CD8, anti CD4, anti CD56 (uterine NK cells), anti FoxP3 primary antibodies will be performed on serial cuts of formalin fixed and paraffin embedded specimens from patients treated with avelumab.
Phenotype of the peritumoral immune cell infiltrate | up to 7 months
  Immunohistochemistry with anti PD-L1, anti CD3, anti CD8, anti CD4, anti CD56 (uterine NK cells), anti FoxP3 primary antibodies will be performed on serial cuts of formalin fixed and paraffin embedded specimens from patients treated with avelumab.

CONTACTS AND LOCATIONS:
Overall Officials: Benoit YOU, MD, Principal Investigator — Hospices Civils de Lyon - Centre Hospitalier Lyon Sud - Service d'Oncologie Médicale
Locations (6):
- France (6):
  - Institut Bergonie, Bordeaux
  - Centre Francois Baclesse, Caen
  - Institut Paoli-Calmettes, Marseille
  - Aphp Hopital Tenon, Paris
  - Hospices Civils de Lyon - CHLS, Pierre-Bénite
  - Institut Universitaire Du Cancer de Toulouse - Oncopole, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] You B, Bolze PA, Lotz JP, Massardier J, Gladieff L, Joly F, Hajri T, Maucort-Boulch D, Bin S, Rousset P, Devouassoux-Shisheboran M, Roux A, Alves-Ferreira M, Grazziotin-Soares D, Langlois-Jacques C, Mercier C, Villeneuve L, Freyer G, Golfier F. Avelumab in Patients With Gestational Trophoblastic Tumors With Resistance to Single-Agent Chemotherapy: Cohort A of the TROPHIMMUN Phase II Trial. J Clin Oncol. 2020 Sep 20;38(27):3129-3137. doi: 10.1200/JCO.20.00803. Epub 2020 Jul 27. PMID 32716740
- [Result] You B, Bolze PA, Lotz JP, Massardier J, Gladieff L, Floquet A, Hajri T, Descargues P, Langlois-Jacques C, Bin S, Villeneuve L, Roux A, Alves-Ferreira M, Grazziotin-Soares D, Dherret G, Gerentet C, Rousset P, Freyer G, Golfier F. Avelumab in patients with gestational trophoblastic tumors with resistance to polychemotherapy: Cohort B of the TROPHIMMUN phase 2 trial. Gynecol Oncol. 2023 Jan;168:62-67. doi: 10.1016/j.ygyno.2022.11.005. Epub 2022 Nov 16. PMID 36401942